CLINICAL TRIAL: NCT01793155
Title: Respiratory Muscle Strength, Functional Capacity and Subjective Outcome - Effects of Inspiratory Muscle Training After Lung Cancer Surgery, a Randomized Controlled Trial
Brief Title: Effects of Inspiratory Muscle Training After Lung Cancer Surgery, a Randomized Controlled Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Region Örebro County (Other); Örebro University, Sweden (Other); KU Leuven (Other)
Responsible Party: Principal Investigator, Barbara C. Brocki, Specialist physiotherapist, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAUH 01; N-201220027 (Other: The Research Ethics Committee in Denmark)
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Lung Cancer; Surgery
Keywords: Lung cancer surgery; Inspiratory muscle training; Postoperative pulmonary complications; Functional outcomes; Health related quality of life
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inspiratory muscle training (Experimental): Inspiratory muscle training for two weeks following surgery
  Interventions: Other: Inspiratory muscle training; Other: Placebo comparator: standard physiotherapy
- Standard physiotherapy (Placebo Comparator): Breathing exercises, cough/hugh, advice on early and active mobilization
  Interventions: Other: Placebo comparator: standard physiotherapy

INTERVENTIONS:
Other: Inspiratory muscle training — Inspiratory muscle training, as a supplement to placebo comparator, starts the day before surgery and continues for two weeks after surgery. No sessions are performed on the surgery day. Each session consists of 2 sets of 30 inspirations with a pause between each set of 2 minutes. The target intensity before surgery is 30% of the measured MIP and starts at 15% after surgery. The intensity is incrementally increased by 2 cm H20 the first days after surgery. Patients grade their perceived exertion and register eventual adverse effects in a training diary.
  Other Names: IMT
  Arms: Inspiratory muscle training
Other: Placebo comparator: standard physiotherapy — Standard physiotherapy - preoperative instruction and postoperative breathing exercises using positive expiratory pressure device (PEP) 3x10 breathings hourly during daytime, cough/huff for mucus clearance purpose, advice on early and active mobilization

SUMMARY:
The purpose of this study is to evaluate the effects of postoperative inspiratory muscle training on the recovery of respiratory muscle strength in high risk patients referred for lung cancer surgery. Furthermore, to assess longitudinal changes in respiratory muscle strength, physical capacity and health-related quality of life after lung cancer surgery

DETAILED DESCRIPTION:
Advances in early detection and treatment improve life expectancy after surgery for lung cancer, but living with lung cancer is frequently associated with symptoms as dyspnoea, decreased physical capacity and fatigue several years after treatment. Lung cancer (LC) surgery is associated with a high incidence of postoperative pulmonary complications (PPC), having a negative impact on recovery. Although the causes of PPC are multifactorial, respiratory muscle (RM) dysfunction has been proposed to be associated with the development of PPC, explained by changes in RM mechanics- and function due to surgery. There is scarcity of literature on the impact of RM dysfunction on surgical and functional outcomes after LC surgery.

Aims: to describe longitudinal changes in RM strength in patients undergoing lung cancer surgery and identify associations between RM strength and functional capacity. Furthermore, to evaluate the effect of inspiratory muscle training on the recovery of respiratory muscle strength in high risk patients referred for LC surgery.

Target population: 88 patients referred for lung cancer surgery at the Department of Cardiothoracic Surgery, Aalborg Universityhospital.

Design: The core of this research is a prospective longitudinal observational study (study 1); included is a randomized controlled trial, based on a subpopulation from study 1.

Statistical analysis is based on mixed linear regression models and ANOVA. For the RCT we use the generalized estimating equivalent method for parametric and Fisher´s exact test for nonparametric data.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years; scheduled for thoracic surgery on the suspicion/confirmed lung tumor via open thoracotomy or Visual Assisted Thoracotomy(includes primary lung cancer, metastases from other cancer sites without activity within none year, other tumor types requiring resection of lung tissue; Furthermore, for RCT, one of the following: Age ≥ 70 years or FEV1 ≤ 70% predicted or DLCO ≤ 70% predicted or scheduled pneumonectomy)

Exclusion Criteria:

* physical or mental deficits that adversely influence physical performance; can neither speak nor read Danish; previous ipsilateral lung resection; tumor activity in other sites or organs; pancoast tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-11; Primary Completion 2014-04 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in inspiratory muscle strength | Before surgery, 5.postoperative day, 2 weeks after surgery
  Change from baseline to 5th postoperative day Change from baseline to 2 weeks after surgery

SECONDARY OUTCOMES:
Change in expiratory muscle strength | Before surgery, 5 th postoperative day and 2 weeks after surgery
  Change from baseline to 5th postoperative day Change from baseline to 2 weeks after surgery
Incidence of postoperative pulmonary complications | 2 weeks after surgery

OTHER OUTCOMES:
Change in walking distance, 6 minute | before surgery, 5th postoperative day and 2 weeks after surgery
  Change from baseline to 5th postoperative day Change from baseline to 2 weeks after surgery
Change in spirometry values(FVC, FEV1) | before surgery, 5th day, 2 weeks after surgery
  Change from baseline to 5th postoperative day Change from baseline to 2 weeks after surgery
Change in Borg CR-10 dyspnea | Before surgery, 5th postoperative day and 2 weeks after surgery
  Change from baseline to 5th postoperative day Change from baseline to 2 weeks after surgery
Change in EORTC QLQ-C30-LC13 | Before surgery and 2 weeks after surgery
Change in EQ-5D-5L | Before surgery and 2 weeks after surgery
Change in Physical Activity Score- PAS | Before surgery and 2 weeks after surgery
Change in numeric rang score for pain | Before surgery, 5th postoperative day and 2 weeks after surgery
  Change from baseline to 5th postoperative day Change from baseline to 2 weeks after surgery
Change in numeric rang score for cough efficiency | 5th postoperative day and 2 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Barbara C Brocki, PT, Principal Investigator — Department of Occupational Therapy- and Physiotherapy, Aalborg Universityhospital
Locations (1):
- Department of Cardiothoracic Surgery, Aalborg Universityhospital, Aalborg, Denmark

REFERENCES:
- [Derived] Brocki BC, Andreasen JJ, Langer D, Souza DS, Westerdahl E. Postoperative inspiratory muscle training in addition to breathing exercises and early mobilization improves oxygenation in high-risk patients after lung cancer surgery: a randomized controlled trial. Eur J Cardiothorac Surg. 2016 May;49(5):1483-91. doi: 10.1093/ejcts/ezv359. Epub 2015 Oct 20. PMID 26489835